CLINICAL TRIAL: NCT06153160
Title: "The Effect of the Use of an Autotransfusion HemaShock Device on Hemodynamic Parameters During Resuscitation"
Brief Title: "The Effect of the Use of an Autotransfusion Device on Hemodynamic Parameters During Resuscitation".
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Collaborators: OHK Medical Devices (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HemaShock socks
Record Dates: First submitted 2023-02-28; First posted 2023-12-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Out of Hospital Cardiac Arrest; Cardiac Arrest
Keywords: Cardiac Arrest; Out of Hospital Cardiac Arrest; Resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with HemaShock device (Experimental): 12 patients in cardiac arrest will receive HemaShock device during resuscitation.
  All other interventions will be made following guidelines.
  Interventions: Device: HemaShock device
- Patients with-out HemaShock device (No Intervention): 12 patients in cardiac arrest will not receive HemaShock device during resuscitation.
  All other interventions will be made following guidelines.

INTERVENTIONS:
Device: HemaShock device — The HemaShock is a tight silicone ring attached to a pressure stocking. It comes wrapped into a doughnut and has a set of handles. The operator simply puts the doughnut over the foot or hand, and pulls on the handles to unravel the HemaShock while applying pressure throughout the appendage. The device displace blood from limbs to central blood system, thus improving preload and cardiac output.
  Arms: Patients with HemaShock device

SUMMARY:
The purpose of the research (pilot study) is to determine the impact of the use of the autotransfusion device on hemodynamic parameters during resuscitation.

24 people will be included in the pilot study (12 people will be included in the intervention group - with the usage of "autotransfusion socks" during resuscitation and 12 people in the control group - without "autotransfusion socks"). Investigators will compare the hemodynamic parameters and also neurological outcome between both groups.

DETAILED DESCRIPTION:
The purpose of the research (pilot study) is to determine the impact of the use of the autotransfusion device on hemodynamic parameters during resuscitation.

Out-of-hospital cardiac arrest (OHCA) is one of the leading causes of death in Europe.

In order to improve the hemodynamic parameters during resuscitation, device for autotransfusion was developed. Devices are basically a very strong elastic stockings that also block arterial circulation. While "putting on" stockings, blood is being squeezed from the lower extremities (approximately 500 ml of blood for each lower limb). With blood being squeezed from the lower limb into the central circulation the filling of the heart is being improved; thus the device will improve the preload and also cardiac output.

A study done on an animal model showed that during resuscitation using "autotransfusion socks" increases both systolic and diastolic blood pressure during resuscitation, the perfusion of the coronary arteries improves and also the values of the partial pressure of carbon dioxide increases.

ELIGIBILITY:
Inclusion Criteria:

* OHCA (Out of Hospital Cardiac Arrest)
* age > 18 years
* intubated
* meets criteria for resuscitation

Exclusion Criteria:

* age < 18 years
* not intubated
* clinical signs for DVT (deep vein thrombosis), PE (pulmonary embolism)
* clinical signs of acute inflammation of limbs, broken limbs etc.
* known oncological patient
* asphyxia
* trauma patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Immediately after arrival to the victim
  Non-invasive blood pressure (both systolic and diastolic blood pressure) will be measured.
End tidal CO2 (Carbon dioxide) after intubation | Immediately after an intubation
  capnography
End tidal CO2 (Carbon dioxide) after application of Hemashock Socks | Immediately after an application of Hemashock Socks
  capnography
End tidal CO2 (Carbon dioxide) every 5 minutes after first application of Hemashock Socks | 5 minutes after the first application of HemaShock socks
  capnography
End tidal CO2 (Carbon dioxide) every 5 minutes after first application of Hemashock Socks | 10 minutes after the first application of HemaShock socks
  capnography
End tidal CO2 (Carbon dioxide) every 5 minutes after first application of Hemashock Socks | 15 minutes after the first application of HemaShock socks
  capnography
End tidal CO2 (Carbon dioxide) every 5 minutes after first application of Hemashock Socks | 20 minutes after the first application of HemaShock socks
  capnography
End tidal CO2 (Carbon dioxide) every 5 minutes after first application of Hemashock Socks | 25 minutes after the first application of HemaShock socks
  capnography
End tidal CO2 (Carbon dioxide) every 5 minutes after first application of Hemashock Socks | 30 minutes after the first application of HemaShock socks
  capnography
End tidal CO2 (Carbon dioxide) after removal of HemaShock Socks | Immediately after the removal of HemaShock socks
  capnography
Blood pressure | Immediately after ROSC
  Noninvasive blood pressure ((both systolic and diastolic blood pressure)) after removal of HemaShock Socks

SECONDARY OUTCOMES:
Cerebral Performance Category Scale | Through study completion, an average of 1 year
  Neurological outcome assessed with Cerebral Performance Category Scale (CPC). CPC 1-2 means good outcome, CPC 3-5 means poor outcome.
Tissue/skin malfunction under HemaShock Socks | From removal of the HemaShock socks up to 15 weeks
  Irrigation, oedema, tissue malperfusion

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Maribor University Medical Centre, Maribor, Maribor City Municipality
  - Community health center Maribor, Prehospital unit, Maribor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyce LW, Vliet Vlieland TP, Bosch J, Wolterbeek R, Volker G, van Exel HJ, Heringhaus C, Schalij MJ, Goossens PH. High survival rate of 43% in out-of-hospital cardiac arrest patients in an optimised chain of survival. Neth Heart J. 2015 Jan;23(1):20-5. doi: 10.1007/s12471-014-0617-x. PMID 25326102
- [Background] Olasveengen TM, Semeraro F, Ristagno G, Castren M, Handley A, Kuzovlev A, Monsieurs KG, Raffay V, Smyth M, Soar J, Svavarsdottir H, Perkins GD. European Resuscitation Council Guidelines 2021: Basic Life Support. Resuscitation. 2021 Apr;161:98-114. doi: 10.1016/j.resuscitation.2021.02.009. Epub 2021 Mar 24. PMID 33773835
- [Background] Soar J, Bottiger BW, Carli P, Couper K, Deakin CD, Djarv T, Lott C, Olasveengen T, Paal P, Pellis T, Perkins GD, Sandroni C, Nolan JP. European Resuscitation Council Guidelines 2021: Adult advanced life support. Resuscitation. 2021 Apr;161:115-151. doi: 10.1016/j.resuscitation.2021.02.010. Epub 2021 Mar 24. PMID 33773825
- [Background] Aminiahidashti H, Shafiee S, Zamani Kiasari A, Sazgar M. Applications of End-Tidal Carbon Dioxide (ETCO2) Monitoring in Emergency Department; a Narrative Review. Emerg (Tehran). 2018;6(1):e5. Epub 2018 Jan 15. PMID 29503830
- [Background] Yang Z, Tang D, Wu X, Hu X, Xu J, Qian J, Yang M, Tang W. A tourniquet assisted cardiopulmonary resuscitation augments myocardial perfusion in a porcine model of cardiac arrest. Resuscitation. 2015 Jan;86:49-53. doi: 10.1016/j.resuscitation.2014.10.009. Epub 2014 Oct 23. PMID 25447436